CLINICAL TRIAL: NCT02124889
Title: Adherence to Multivitamin Use Following Bariatric Surgery for Weight Loss
Brief Title: Multivitamin Adherence Following Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Celebrate Vitamins (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00027050
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: bariatric surgery; multivitamin; weight loss; adherence
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either receive the weekly survey or not.
Who Masked: Investigator
Masking Description: The Pi does not know which participants are randomized to get the weekly survey.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly surveys (Experimental): Subjects will take the multivitamin, and will also receive weekly Internet surveys asking them questions about the multivitamin treatment.
  Interventions: Behavioral: Weekly Internet surveys
- No Survey (No Intervention): Subjects will take the multivitamin.

INTERVENTIONS:
Behavioral: Weekly Internet surveys — Subjects will receive weekly Internet surveys asking them how their treatment is working, how often they took the medication, and how easy it was to use the medication.
  Arms: Weekly surveys

SUMMARY:
Additional micronutrient supplementation is required due to the changes in the gastrointestinal anatomy and physiology following bariatric surgery along with decreased dietary intake and rapid weight loss. Good adherence to post-operative vitamins is essential to maintain healthy vitamin levels in the body following bariatric surgery. The hypothesis of this study is that patients receiving a weekly survey intervention will have better adherence to post-operative vitamins.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo a Roux En Y Gastric Bypass or Sleeve Gastrectomy at Wake Forest Baptist Health

Exclusion Criteria:

* Admission for a psychiatric event in the past year
* History of nausea and/or significant complaint of post-operative nausea
* History of stricture and/or significant complaint of post-operative stricture
* History of ulcer and/or significant complaint of post-operative ulcer
* History of major depression or psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Z Fernandez, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Weekly Surveys: Subjects will take the multivitamin, and will also receive weekly Internet surveys asking them questions about the multivitamin treatment.
  Weekly Internet surveys: Subjects in this arm will receive weekly Internet surveys asking them how their treatment is working, how often they took the medication, and how easy it was to use the medication.
- No Survey: Group will only get multivitamin - no weekly survey
Period: Overall Study
Arm/Group | Weekly Surveys | No Survey
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Survey - Control: Subjects will take the multivitamin but will not receive surveys.
- Total: Total of all reporting groups
Arm/Group | Weekly Surveys | No Survey - Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Multivitamin
Description: Percent of anticipated number of doses the patient has taken, as recorded by a Medication Event Monitoring System (MEMS) cap.
Time Frame: 50 days
Measure: Mean (Standard Error); unit: percentage of doses taken
Arm/Group | Weekly Surveys | No Survey
Number analyzed (Participants) | 12 | 12
percentage of doses taken | 32.9 (5.93) | 34.9 (5.91)

ADVERSE EVENTS:
Groups:
- No Survey - Control: Subjects will take the multivitamin without additional contact.
Arm/Group | Weekly Surveys | No Survey - Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No